CLINICAL TRIAL: NCT02179255
Title: An Open-Label Randomized Controlled Trial (RCT) of 6 Weeks of Human Growth Hormone (HGH) Prior to Ovulation Induction for In Vitro Fertilization (IVF)
Brief Title: Human Growth Hormone Pre-treatment for 6 Weeks Prior to Ovulation Induction for IVF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04082014-02
Record Dates: First submitted 2014-06-15; First posted 2014-07-01 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve
Keywords: DOR; Premature Ovarian Failure (POF); Ovarian Failure; Human Growth Hormone
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Human Growth Hormone; Growth Hormone; Follicle Stimulating Hormone; Urofollitropin; follitropin beta; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Growth Hormone (Experimental): 1.9 mg (5.7 units) daily injection of Recombinant Human Growth Hormone (HGH) for at least 6 weeks (42 days) plus FSH 450 to 600 units per day administered subcutaneous (SQ) daily dose adjusted based on the patients response starting on day 2 of the 28 day menstrual cycle and continued until Ovulation trigger
  Interventions: Drug: Human Growth Hormone; Drug: Follicle Stimulating Hormone
- Follicle Stimulating Hormone (Active Comparator): FSH 450 to 600 units per day administered SQ daily dose adjusted based on the patients response starting on day 2 of the 28 day menstrual cycle and continued until Ovulation trigger
  Interventions: Drug: Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Human Growth Hormone — 1.9 mg (5.7 units) daily injection of Recombinant Human Growth Hormone (HGH) for at least 6 weeks (42 days) continuing into the approximately 14 days of ovulation induction phase of the trial.
  Other Names: Human Growth Hormone (HGH); Somatotropin; Omnitrope; Norditropin; Humatrope; Saizen; Genotropin; Serostim; Nutropin; Tev-tropin; Zorbtive
  Arms: Human Growth Hormone
Drug: Follicle Stimulating Hormone — FSH 450 to 600 units per day administered SQ daily dose adjusted based on the patients response starting on day 2 of the 28 day menstrual cycle and continued until Ovulation trigger
  Other Names: Bravelle; Follistim; Gonal-F; Menopure

SUMMARY:
Synthetic human growth hormone (HGH) has been available for more than a decade for specific indication in children and adults. Past Randomized Control Trials (RCT)s of HGH (under off-label use) for improving ovarian function have shown that a combination of traditional gonadotropin ovulation induction protocols, with addition of HGH is effective in increasing pregnancy rates, but not increasing egg production after IVF in women with documented diminished ovarian reserve (DOR). The investigators hypothesize that by initiating HGH at least 6 weeks prior to IVF start, the investigators will be able to increase production of oocytes and further improve pregnancy chances. This hypothesis is based on prior observations of effects of growth hormone on small antral follicles and the fact that prior studies utilized HGH principally only during ovulation induction itself.

The investigators plan to recruit 30 women (15 in each group) to an open label randomized controlled trial of HGH for augmentation of ovarian response among women with documented DOR and poor prior response to ovulation induction.

Eligible participants will be women < 45 years with documented history of prior retrieval of 2 or fewer oocytes while on maximal ovulation induction despite prior supplementation with dehydroepiandrosterone (DHEA).

Women will be treated with 1.9 mg (5.7 units) of HGH per day, beginning about 6 weeks before start of their treatment cycle. Cost of treatment with HGH will be a cost to the participating patient. HGH will cost the patient approximately $800 per week of treatment. Patients who are randomized to the non-HGH treated group, and do not conceive, will in the following cycle be offered HGH supplementation outside of this clinical trial. This subsequent cycle will not be part of the study dataset and patients will also be responsible for the cost of HGH.

Even with only 7 patients in each group, this trial will have a 99% power (error 0.05%) to detect a mean increase to 4 oocytes in the treated group. The investigators plan to recruit 15 patients in each group to allow for possible dropouts.

DETAILED DESCRIPTION:
Synthetic HGH was developed in 1985 and approved by the FDA for specific uses in children and adults (1996; 2003). In children, HGH injections are approved for treating short stature of unknown cause as well as poor growth due to a number of medical causes, including:

* Turner's syndrome, a genetic disorder that affects a girl's development.
* Prader-Willi syndrome, an uncommon genetic disorder causing poor muscle tone, low levels of sex hormones, and a constant feeling of hunger.
* Chronic kidney insufficiency.
* HGH deficiency or insufficiency.
* Children born small for gestational age.

In adults, approved uses of HGH include:

* Short bowel syndrome, a condition in which nutrients are not properly absorbed due to severe intestinal disease or the surgical removal of a large portion of the small intestine.
* HGH deficiency due to rare pituitary tumors or their treatment.
* Muscle-wasting disease associated with HIV/AIDS.

HGH supplementation is potentially useful in ovulation induction. Over the last decade, as recombinant HGH has become commercially available, there have been many studies looking at the effects of HGH on ovulation induction. Almost all of these studies administered HGH along with routine fertility medication during the ovulation induction cycle. Most studies used HGH doses between 4 units and 12 Units. A few studies started GH on day 21 of the previous cycle.

A recent Cochrane review found that, while HGH did not improve results in routine IVF cycles there is "some evidence of increased pregnancy and birth rates in women who are considered 'poor responders' to in vitro fertilization."

HGH is reported to modulate the action of follicle stimulating hormone (FSH) on follicles by up-regulating local synthesis of IGF-1. A similar effect was, interestingly, noted by Casson et al. (Casson, Santoro et al. 1998; Casson, Lindsay et al. 2000) in early experiments using DHEA with treated patients having increased IGF-1. Much of the focus on gonadotropin /IGF-1

interaction has revolved around the effects on granulosa cell cultures to increase aromatase activity, estradiol production progesterone production and Luteinizing Hormone (LH) receptor formation. However,Insulin-Like Growth Factor-1 (IGF-1) also has a proposed role in stimulating early follicle development and oocyte maturation (Yoshimura, Ando et al. 1996; Yoshimura, Aoki et al. 1996).

Based on these observations, we believe that HGH in past trials has not been used to maximal effect. Since HGH, like DHEA, appears to affect small growing follicles, weeks to months removed from gonadotropin sensitivity, the greatest potential for HGH, under our hypothesis, would be its use, attempting to affect these small growing follicles. In analogy to DHEA supplementation, this would mean that HGH supplementation would have to be initiated at least 6 weeks prior to IVF cycle stimulation start. Theoretically, administration of HGH during the 6 week before starting an IVF cycle will have an effect on developing antral follicles to present a larger and better quality cohort of follicles when ovulation induction is begun.

ELIGIBILITY:
Inclusion Criteria:

* The study will be limited to women with Poor Response to prior treatment with evidence of diminished ovarian reserve with 2 or fewer oocytes in a previous ovulation induction cycles with maximal gonadotrophin stimulation. All women in this study will be <45 years old.

Exclusion Criteria:

* Cardiac disease, evidence of glucose intolerance

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Oocytes retrieved for IVF | 8 weeks after starting intervention

SECONDARY OUTCOMES:
Clinical Pregnancy Rates | 12 weeks after starting intervention
  Presence of an established clinical pregnancy as evidenced by gestational sac with active fetal heart beat

CONTACTS AND LOCATIONS:
Overall Officials: David H Barad, MD, Principal Investigator — Center for Human Reproduction; Norbert Gleicher, Study Chair — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

REFERENCES:
- [Background] FDA approves human growth hormone for wasting syndrome. AIDS Patient Care STDS. 1996 Dec;10(6):379-80. No abstract available. PMID 11361571
- [Background] FDA approves growth hormone for short children. Child Health Alert. 2003 Sep;21:4. No abstract available. PMID 14552287
- [Background] Bergh C, Hillensjo T, Wikland M, Nilsson L, Borg G, Hamberger L. Adjuvant growth hormone treatment during in vitro fertilization: a randomized, placebo-controlled study. Fertil Steril. 1994 Jul;62(1):113-20. PMID 7516295
- [Background] Dor J, Seidman DS, Amudai E, Bider D, Levran D, Mashiach S. Adjuvant growth hormone therapy in poor responders to in-vitro fertilization: a prospective randomized placebo-controlled double-blind study. Hum Reprod. 1995 Jan;10(1):40-3. doi: 10.1093/humrep/10.1.40. PMID 7745068
- [Background] Suikkari A, MacLachlan V, Koistinen R, Seppala M, Healy D. Double-blind placebo controlled study: human biosynthetic growth hormone for assisted reproductive technology. Fertil Steril. 1996 Apr;65(4):800-5. doi: 10.1016/s0015-0282(16)58217-x. PMID 8654642
- [Background] Bergh C, Carlstrom K, Selleskog U, Hillensjo T. Effect of growth hormone on follicular fluid androgen levels in patients treated with gonadotropins before in vitro fertilization. Eur J Endocrinol. 1996 Feb;134(2):190-6. doi: 10.1530/eje.0.1340190. PMID 8630518
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- [Background] Casson PR, Santoro N, Elkind-Hirsch K, Carson SA, Hornsby PJ, Abraham G, Buster JE. Postmenopausal dehydroepiandrosterone administration increases free insulin-like growth factor-I and decreases high-density lipoprotein: a six-month trial. Fertil Steril. 1998 Jul;70(1):107-10. doi: 10.1016/s0015-0282(98)00121-6. PMID 9660430
- [Background] Hazout A, Junca Am, Menezo Y, Demouzon J, Cohen-Bacrie P. Effect of growth hormone on oocyte competence in patients with multiple IVF failures. Reprod Biomed Online. 2009 May;18(5):664-70. doi: 10.1016/s1472-6483(10)60011-9. PMID 19549445
- [Background] Kucuk T, Kozinoglu H, Kaba A. Growth hormone co-treatment within a GnRH agonist long protocol in patients with poor ovarian response: a prospective, randomized, clinical trial. J Assist Reprod Genet. 2008 Apr;25(4):123-7. doi: 10.1007/s10815-008-9212-7. PMID 18392675
- [Background] Owen EJ, Shoham Z, Mason BA, Ostergaard H, Jacobs HS. Cotreatment with growth hormone, after pituitary suppression, for ovarian stimulation in in vitro fertilization: a randomized, double-blind, placebo-control trial. Fertil Steril. 1991 Dec;56(6):1104-10. doi: 10.1016/s0015-0282(16)54724-4. PMID 1743329
- [Background] Tesarik J, Hazout A, Mendoza C. Improvement of delivery and live birth rates after ICSI in women aged >40 years by ovarian co-stimulation with growth hormone. Hum Reprod. 2005 Sep;20(9):2536-41. doi: 10.1093/humrep/dei066. Epub 2005 Apr 28. PMID 15860489
- [Background] Yoshimura Y, Ando M, Nagamatsu S, Iwashita M, Adachi T, Sueoka K, Miyazaki T, Kuji N, Tanaka M. Effects of insulin-like growth factor-I on follicle growth, oocyte maturation, and ovarian steroidogenesis and plasminogen activator activity in the rabbit. Biol Reprod. 1996 Jul;55(1):152-60. doi: 10.1095/biolreprod55.1.152. PMID 8793070
- [Background] Demeestere I, Gervy C, Centner J, Devreker F, Englert Y, Delbaere A. Effect of insulin-like growth factor-I during preantral follicular culture on steroidogenesis, in vitro oocyte maturation, and embryo development in mice. Biol Reprod. 2004 Jun;70(6):1664-9. doi: 10.1095/biolreprod.103.023317. Epub 2004 Feb 11. PMID 14960488
- [Background] Yoshimura Y, Aoki N, Sueoka K, Miyazaki T, Kuji N, Tanaka M, Kobayashi T. Interactions between insulin-like growth factor-I (IGF-I) and the renin-angiotensin system in follicular growth and ovulation. J Clin Invest. 1996 Jul 15;98(2):308-16. doi: 10.1172/JCI118794. PMID 8755639
- [Background] Zhuang GL, Wong SX, Zhou CQ. [The effect of co-administration of low dosage growth hormone and gonadotropin for ovarian hyperstimulation in vitro fertilization and embryo transfer]. Zhonghua Fu Chan Ke Za Zhi. 1994 Aug;29(8):471-4, 510. Chinese. PMID 7835118
- [Derived] Sood A, Mohiyiddeen G, Ahmad G, Fitzgerald C, Watson A, Mohiyiddeen L. Growth hormone for in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD000099. doi: 10.1002/14651858.CD000099.pub4. PMID 34808697